CLINICAL TRIAL: NCT05755152
Title: Fruit-based Chewing Gums for Improving Oral Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Wisconsin Alumni Research Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2022-1703; Protocol Version 1/12/2023 (Other: UW Madison); Food Science (Other: UW Madison); Discovery 2 Product (Other: UW Madison)
Record Dates: First submitted 2023-02-17; First posted 2023-03-06 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Oral Health
Keywords: Cranberry; Bioavailability; Polyphenol

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to their first intervention and cross over to the second intervention.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cranberry PLP (Experimental): Chew the treatment chewing gum made with PLP at specific time intervals for a total of 60 minutes
  Interventions: Other: polyphenol-lecithin precipitate (PLP)
- Cranberry Extract Control (Experimental): Chew the control chewing gum made with Cranberry Extract at specific time intervals for a total of 60 minutes
  Interventions: Other: control formulation

INTERVENTIONS:
Other: polyphenol-lecithin precipitate (PLP) — Chewing gum made with material produced from patented technology to rapidly isolate polyphenols from fruit juice (PLP).
  Arms: Cranberry PLP
Other: control formulation — Chewing gum made with material produced from conventional technology (e.g cranberry extract).
  Arms: Cranberry Extract Control

SUMMARY:
This study aims to conduct a randomized cross-over study investigating the release of cranberry polyphenols from chewing gum formulated with polyphenol-lecithin precipitate (PLP). 10 participants will be on study for up to 2 weeks and will each complete 2-30 minute study intervention visits.

DETAILED DESCRIPTION:
This study is intended to evaluate the bioavailability of a dietary supplement, cranberry PLP, compared to another dietary ingredient, cranberry extract. The intent of the evaluation is to provide preliminary data for future evaluation of cranberry PLP on the normal structure or function in humans, which includes the effect of cranberry PLP on oral health.

Participants will be asked to refrain from eating, drinking, or using tobacco products, and vigorous exercise for 1 hour before the intervention period. Participants will also be asked to avoid chewing gum 48 hours before the intervention. Water is acceptable up until 10 minutes before sample collection. Participants will be given these instructions during the informed consent process, and will be sent a reminder email about study protocols at least 72 hours in advance of the study visit. If their second visit is 48 hours after their first, the investigators will remind them of these restrictions at the end of their first visit.

On the day of each intervention and sampling period, participants will be asked to visit the Bolling Laboratory at the Department of Food Science adhering to the dietary guidance described above. Participants with appliances or dentures will be asked to remove them during sampling periods. Then, participants will chew the intervention or control gum for a total of 60 minutes while providing chewed gum and saliva samples at specified intervals throughout this time. Participants will come back to the Bolling Laboratory at a later time, a minimum of 48 hours after the last sampling period, to chew the other gum in the same manner as the first sampling period.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults 18 years and older
* willing to avoid foods, beverages, tobacco products, and additional gum in the wash-in and wash-out periods
* willing to chew the intervention gum during the sampling periods
* willing to provide saliva and gum samples during the sampling periods
* willing to fill out post-visit surveys after their visits

Exclusion Criteria:

* Participants who do not consider themselves healthy
* have less than 20 natural teeth and 8 natural posterior teeth (excluding third molars)
* have a salivary rate ≥ 0.3 mL/min as determined from an unstimulated salivary flow trial
* taking medications that contraindicates grapefruit juice consumption
* allergic to any intervention foods or ingredients (e.g. sunflower, soy, food colorants, berry ingredients, or any other component of the study gum)
* diagnosed with phenylketonuria (PKU), gross untreated caries, advanced gingivitis and periodontitis, and temporomandibular joint disorder
* participants who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2023-10-26 (Actual)

PRIMARY OUTCOMES:
Concentration of Polyphenols | Baseline before chewing gum; then 1, 3, 6, 10, 15, 21 minutes after start of chewing gum.
  Participant chewed gum samples will be measured for polyphenol concentration.

SECONDARY OUTCOMES:
pH | Baseline before chewing gum and approximately 60 minutes after start of chewing gum.
  Participant saliva samples will be measured for pH.
Concentration of Polyphenols | Baseline before chewing gum and approximately 60 minutes after start of chewing gum.
  Participant saliva samples will be measured for polyphenol concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Bolling, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Babcock Hall, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-03-07): https://cdn.clinicaltrials.gov/large-docs/52/NCT05755152/ICF_000.pdf